CLINICAL TRIAL: NCT04296253
Title: Angiogenic Growth Factors, Pro- and Anti-inflammatory Biomarkers, and Genetic Polymorphisms of Their Promoter Regions in Patients With Post-infarction Cardiac Remodeling
Brief Title: Biomarkers and SNP-polymorphisms in Post-infarction Cardiac Remodeling
Status: Completed | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Vyacheslav Ryabov, Deputy Director for Research and Clinical Services of Cardiology Research Institute, Head of Department of Emergency Cardiology, Clinical Professor, Principal Invastigator, Tomsk National Research Medical Center of the Russian Academy of Sciences
Other Study IDs: SNP_1
Record Dates: First submitted 2019-03-31; First posted 2020-03-05 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Myocardial Infarction
Keywords: remodeling; inflammation; polymorphism; endotoxin; heart failure
MeSH Terms: conditions — Myocardial Infarction; Inflammation; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be obtained from patients with acute ST segment elevation myocardial infarction, who underwent coronary angiography within 24 hours of the onset of the disease.

INTERVENTIONS:
Genetic: SNP polymorphisms of the promoter regions pro - and anti-inflammatory cytokines and angiogenic growth factor — blood sampling

SUMMARY:
The purpose of this study is to explore the serum levels of pro- and anti-inflammatory biomarkers and angiogenic growth factors and SNP polymorphisms of the promoter regions of their genes as well as to determine their role in the development of adverse cardiac remodeling in patients with acute ST-segment elevation myocardial infarction.

DETAILED DESCRIPTION:
The widespread introduction of modern methods of treatments of myocardial infarction in routine clinical practice has lead not only to a decrease in mortality, but also to an increase in the number of patients with chronic heart failure. It is known that inflammation develops in myocardial infarction in response to cell damage, which is accompanied by activation of the cells of the immune system and eventually with scarring. Chronic aseptic inflammation is not only a universal biological reaction in response to necrosis of cardiomyocytes, but the cellular molecular basis of post-infarction cardiac remodeling. At the same time, the imbalance of pro- and anti-inflammatory mediators can have some negative effects on the healing processes of the damaged myocardium and subsequent remodeling of the heart. In adverse heart remodeling, elevated levels of proinflammatory cytokines (IL-1β, IL-6, TNF-α, etc.) and reduced secretion of anti-inflammatory cytokines (IL-4, IL-10, etc.) persist for a long time.

Recently, the endotoxin hypothesis of cytokine production has been of great interest among scientists. Endotoxin is a molecule of the lipopolysaccharide (LPS) of the outer cell wall of gram-negative bacteria. LPS is a powerful inducer of cytokine release, and chronic endotoxin load is at least one of the reasons for the activation of the innate immune system. One of the most important and unresolved problems in pathophysiology is the study of the nature of the inflammatory response, or rather the cytokine response cascade, reparation and neoangiogenesis developing in the myocardium in response to ischemic damage, as well as genetically determined regulation of these processes. Factors determining the dual role of cytokines in the development of adverse cardiac remodeling can be polymorphisms of their genes, in particular, single nucleotide polymorphism of genes - SNP (single nucleotide polymorphism) with replacement of one nucleotide by another. SNP in promoter regions regulate the intensity of gene expression, different levels of secretion and function of interleukins, growth factors, and, accordingly, their biological effects. Uncovering the mechanisms that regulate the secretion of angiogenic growths factors, pro- and anti-inflammatory cytokines in patients with AMI could potentially become the basis for developing new treatment tactics based on modulating the immune response and neoangiogenesis in AMI by introducing into ischemic tissues of cytokines or angiogenic growth factors in the form recombinant proteins or as a part of genetic constructs to stimulate regeneration.

A total of 200 patients with acute primary myocardial infarction with ST segment elevation will be recruited. Upon admission, all patients receive standard therapy, as recommended for the treatment of myocardial infarction. Within 24 hours of admission, coronary angiography and revascularization of the infarct-related artery are performed. On the days 1 and 7 of hospitalization and on the day of discharge, blood will be taken to determine the dynamics of serum concentrations of pro- and anti-inflammatory biomarkers, markers of myocardial necrosis; gene polymorphisms will be studied; echocardiography will be performed to assess the structural and functional characteristics of the heart after AMI. After 3 and 12 months, patients undergo studies to dynamically assess the structural and functional state of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of randomization
* Patients with acute coronary syndrome with ST segment elevation
* Signed informed consent to participate in the study
* Admission to the intensive care unit within 24 hours from the onset of the disease
* Coronary angiography within 24 hours of the onset of the disease

Exclusion Criteria:

* Long persistent form of atrial fibrillation
* Valvular heart disease
* Shock of different genesis
* Multiple organ failure
* Chronic heart failure with a severe decrease in the left ventricular ejection fraction
* Sepsis
* Severe concomitant pathology

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction with ST segment elevation, who underwent coronary angiography within 24 hours of the onset of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in the left ventricular end-diastolic volume index (percent) | 1 year
  Change in the left ventricular end-diastolic volume index (percent) is assessed in patients with myocardial infarction at 1-year follow-up with intermediate assessments at day 7 and month 3 after onset.

SECONDARY OUTCOMES:
Incidence of mortality (percent) | 1 year
  Incidence rate of mortality (percent) is measured 1 year after myocardial infarction onset.
Incidence of stroke (percent) | 1 year
  Incidence rate of stroke (percent) is measured 1 year after myocardial infarction onset.
Incidence of unstable angina (percent) | 1 year
  Incidence rate of unstable angina (percent) is measured 1 year after myocardial infarction onset.
Incidence of chronic heart failure > II NYHA (percent) | 1 year
  Incidence rate of chronic heart failure (percent) is measured 1 year after myocardial infarction onset.
Incidence of recurrent myocardial infarction (percent) | 1 year
  Incidence rate of recurrent myocardial infarction (percent) is measured 1 year after myocardial infarction onset.
Change in pro-inflammatory cytokine (pg/mL) | 1 year
  Changes in the serum levels of pro-inflammatory cytokines (pg/mL) in patients with myocardial infarction is assessed at 1-year follow-up with intermediate assessments at days 1, 7 and 14 and month 3 after onset.
Change in anti-inflammatory cytokine (pg/mL) | 1 year
  Changes in the serum levels of anti-inflammatory cytokines (pg/mL) in patients with myocardial infarction is assessed at 1-year follow-up with intermediate assessments at days 1, 7 and 14 and month 3 after onset.
Change in angiogenic growth factor (pg/mL) | 1 year
  Changes in the serum levels of angiogenic growth factors (pg/mL) in patients with myocardial infarction at 1-year follow-up with intermediate assessments at days 1, 7 and 14 and month 3 after onset.
Change in endotoxin (ng/mL) | 1 year
  Changes in the serum levels of endotoxin (ng/mL) in patients with myocardial infarction at 1-year follow-up with intermediate assessments at days 1, 7 and 14 and month 3 after onset.

OTHER OUTCOMES:
CE 1: cardiovascular mortality + myocardial reinfarction + unstable angina (percent) | 1 year
  Combined incidence rate of cardiovascular mortality, myocardial reinfarction, and unstable angina (percent) is measured 1 year after myocardial infarction onset.
CE 2: cardiovascular mortality + myocardial reinfarction + chronic heart failure > II NYHA (percent) | 1 year
  Combined incidence rate of cardiovascular mortality, myocardial reinfarction, and chronic heart failure NYHA functional class III and IV (percent) is measured 1 year after myocardial infarction onset.

CONTACTS AND LOCATIONS:
Overall Officials: Vyacheslav Ryabov, MD, PhD, Principal Investigator — Cardiology Research Institute, Tomsk NRMC
Locations (1):
- Cardiology Research Institute of Tomsk National Research Medical Center of the Russian Academy of Sciences, Tomsk, Tomskii Region, Russia